CLINICAL TRIAL: NCT05625217
Title: Characterizing Dynamics of FDG Uptake With Total-Body PET for Response Assessment in Radiotherapy for Head and Neck Cancer
Brief Title: Total-Body FDG PET for Radiotherapy Response Assessment in Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1946919
Record Dates: First submitted 2022-11-07; First posted 2022-11-22 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Total-body PET scan (Experimental): All participants are asked to complete two study scan visits. First visit occurs before treatment and the second visit occurs 12 +/- 2 weeks after treatment. Each visit will involve a single injection of FDG, followed by three PET/CT scans that will start immediately following injection, at about 2 hours post-injection and at 5 hours post-injection, respectively and last about 60 minutes, 20 minutes and 20 minutes, respectively.
  Interventions: Diagnostic Test: Total Body PET/CT Imagin

INTERVENTIONS:
Diagnostic Test: Total Body PET/CT Imagin — Total-body PET imaging at different timepoints

SUMMARY:
The overall goal of this research study is to understand how 18F-fluorodeoxyglucose (FDG), a radioactive sugar behaves in head and neck cancer (HNC) and inflammation immediately following injection and at many hours post-injection, with the world's first total-body positron emission tomography (PET)/computed tomography (CT) scanner (EXPLORER).

ELIGIBILITY:
Inclusion Criteria:

1. Stage II-IVa (American Joint Committee on Cancer, 8th edition) OC who are planned for RT (≥60 Gy) as per routine clinical standard.
2. Patient must be ≥18 years of age.
3. Willing and able to lay motionless in a supine position for up to 60 minutes
4. Patient must be able to provide study specific informed consent prior to study entry.
5. Patient must be able to adhere to the study visit schedule and other protocol requirements (including prolonged fasting).

Exclusion Criteria:

1. Prior RT for any malignancy leading to overlap with planned RT fields.
2. Prior chemotherapy for any malignancy.
3. Subjects suffering from severe claustrophobia.
4. Subjects who have had a research study involving radiation within one year of enrolling in this study
5. Subjects who are pregnant (subjects 18 to 60 years old who are able to become pregnant unless documented hysterectomy or bilateral ovarian removal is available will be tested prior to injection of imaging agent - positive test will exclude from participating in the study)
6. Subjects who are breastfeeding
7. Prisoners.
8. Any significant medical condition that in the opinion of the investigator would prevent the subject from participating and/or adhering to study related procedures or interfere with subject safety (e.g., poorly controlled diabetes).
9. Children (<18 years of age).
10. Body weight more than 240 kg (529 pounds)

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Utility of long-delayed FDG PET Imaging | Percent change from baseline to 2 hour post injection
  The retention index based on the SUVmax for Oral Cancer and Radiotherapy-induced inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Tokihiro Yamamoto, PhD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis EXPLORER Molecular Imaging Center, Sacramento, California, United States